CLINICAL TRIAL: NCT03015376
Title: Cohort Study on Characters and Distribution of Inherited Susceptible Genes Among Epithelial Ovarian Cancer Patients and Their Relatives in the North of China
Brief Title: Inherited Susceptible Genes Among Epithelial Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, associate professor, Peking Union Medical College Hospital
Other Study IDs: EOC-GENE
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Ovarian Neoplasm Epithelial; Hereditary Breast and Ovarian Cancer Syndrome
Keywords: epithelial ovarian cancer; Hereditary Breast and Ovarian Cancer Syndrome; next-generation sequencing; High-Throughput Nucleotide Sequencing
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum from peripheral blood and tumor tissues frome surgical samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose: To investigate the prevalence of the germline mutations in the BRCA 1/2 and mismatch repair genes in patients with epithelial ovarian cancer (EOC) and their relatives, and related somatic mutations in tumor tissues in the northern part of china.

Patients and methods: A multicenter prospective study will be hold in the northern part of china form 2017. About 1000 female patients with epithelial ovarian cancer and their ralatives will be tested for germline mutations in the BRCA 1/2 and mismatch repair genes and related somatic mutations in tumor tissues, regardless of the family history.

Study type: Observational Official title: Prevalence study of germline mutations in susceptibility ovarian cancer genes in patients with epithelial ovarian cancer and somatic mutations in their tumor tissures in the northern part of china.

Enrollment: 1000

ELIGIBILITY:
Inclusion Criteria:

1. epithelial ovarian cancer and their relatves
2. living in the north of Huaihe River in China
3. being Han Chinese

Exclusion Criteria:

1. non-epithelial ovarian cancer
2. without specific pathological diagnosis
3. non-Han Chinese

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patiens with epithelia ovarian cancer and their relatves in the North of China
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
herited gene mutations susceptible to epithelial ovarian cancer in patients and their relatives | two years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Ming, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Lei Li, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with authorised researchers via online database.

REFERENCES:
- [Derived] Li W, Shao D, Li L, Wu M, Ma S, Tan X, Zhong S, Guo F, Wang Z, Ye M. Germline and somatic mutations of multi-gene panel in Chinese patients with epithelial ovarian cancer: a prospective cohort study. J Ovarian Res. 2019 Aug 31;12(1):80. doi: 10.1186/s13048-019-0560-y. PMID 31472684
- [Derived] Li L, Ma S, Tan X, Zhong S, Wu M. The Urodynamics and Survival Outcomes of Different Methods of Dissecting the Inferior Hypogastric Plexus in Laparoscopic Nerve-Sparing Radical Hysterectomy of Type C: A Randomized Controlled Study. Ann Surg Oncol. 2019 May;26(5):1560-1568. doi: 10.1245/s10434-019-07228-8. Epub 2019 Feb 13. PMID 30759291